CLINICAL TRIAL: NCT03344016
Title: The MUPPET-study: Multicenter Pheochromocytoma and Paraganglioma Evaluation for Follow-up Screening, Genetics Sub-Typing, Therapy and Outcome
Brief Title: Multicenter Pheochromocytoma and Paraganglioma Evaluation
Acronym: MUPPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Felix Beuschlein (Other)
Collaborators: Technische Universität Dresden (Other); Wuerzburg University Hospital (Other); University of Zurich (Other); Radboud University Medical Center (Other); Lübeck University Clinic (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor-Investigator, Felix Beuschlein, Prof., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 742-16
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Intervention Model Description: To provide evidence whether strict follow-up will result in improvement in clinical outcome parameters as compared to standard care follow-up, patients upon inclusion into the study protocol will be randomized into two groups:
  * Standard care follow-up group: Patients will receive an information leaflet (see appendix), which advises on recommended routine follow-up according to international guidelines.
  * Special care follow-up group: In addition to the information leaflet patients will be actively contacted by the clinical center to increase the likelihood that patients meet recommended follow-up schedules.
  Stratification will be done for inclusion criteria (newly diagnosed PPGL, previous history of PPGL, gene carrier, presence of malignant PPGL and center).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care follow-up group (No Intervention): Patients will receive an information leaflet (see appendix), which advises on recommended routine follow-up according to international guidelines.
- Special care follow-up group (Active Comparator): In addition to the information leaflet patients will be actively contacted by the clinical center to increase the likelihood that patients meet recommended follow-up schedules.
  Interventions: Other: Contact by clinical center

INTERVENTIONS:
Other: Contact by clinical center — Patients will be acitvely contacted by the clinical center for follow-up procedure
  Arms: Special care follow-up group

SUMMARY:
Target population:

Patients with (1) newly diagnosed or (2) past history of pheochromocytomas and paragangliomas (PPGL) or (3) carrier of genetic mutations in known PPGL susceptibility genes.

International multicenter prospective cohort study with randomized intervention (special care follow-up vs. standard care follow-up).

All patients will receive instructions about follow-up at the time point of study inclusion. Patients randomized to the standard care follow-up group will be advised to return annually for follow-up according to current routine practice (without active re-scheduling). In contrast, patients randomized to the special care follow-up group will also be advised to return annually for follow-up but these patients will be actively invited, re-scheduled and reminded by the centers to meet scheduled follow-up appointments.

DETAILED DESCRIPTION:
The long-term goal of the research planned under this protocol is to reduce morbidity and mortality of patients with PPGLs by improving approaches for management, follow-up and therapy of affected patients. As a first step towards attaining this goal, the primary objective of this protocol is to investigate whether standardized follow-up results in improved long-term outcome in terms of less morbidity and mortality as compared. The central hypothesis is that pro-active, structured and periodic disease screening and management of patients at risk for developing PPGLs and other neoplasms can lead to earlier detection of tumors and reduce adverse outcomes associated with cardiovascular, metabolic and oncologic complications of the tumors than standard care follow-up. The underlying rationale is that establishing improved outcomes for patients at risk for PPGLs will enable evidence-based recommendations for disease follow-up and management, thereby establishing wider acceptance and use of outlined practices with ensuing improvements in the health and quality of life of affected patients and their families.

In addition to the primary objective directed at establishing whether standardized and structured follow-up of patients with an increased risk for new events of PPGL (recurrent tumor, new tumor, or metastases) will result in improved longterm outcome, this protocol will enable several secondary objectives to be addressed using clinical (e.g. age, mode of presentation), biochemical, metabolic and genetic characteristics. These include:

1. to identify prognostic markers of disease progression
2. to assess whether clinical presentation, cardiovascular, metabolic and biochemical phenotype, genetic background and tumor characteristics (location, size, recurrence, pathology) are useful for development of personalized follow-up strategies.
3. to investigate whether standardized follow-up affects quality of life

ELIGIBILITY:
Inclusion Criteria:

male and female patients (≥ 5 years of age), who fulfill one or more of the following criteria: (i) Patients with a newly diagnosed PPGL. (ii) Patients with a previous history of PPGLs. (iii) Carrier of genetic mutations known to predispose for the development of PPGLs.

All subjects must have read, understood and signed the informed consent form, before inclusion into the study protocol. Signed parental consent must be obtained for children with suspected PPGLs who are enrolled in the study.

Exclusion Criteria:

* Patients with impaired mental capacity that precludes informed consent.
* Pregnancy does not constitute criteria for exclusion from the protocol. However, in pregnant women no Clonidine testing, no PET scanning, MIBG scanning or contrast CT will be performed.
* Patients at risk from injury from the MRI magnet due to implantable metal or who suffer from anxiety in enclosed spaces are excluded from MRI.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1148 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2035-11-01 (Estimated); Study Completion 2040-11-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 18 years
  to investigate whether standardized follow-up for patients at risk for PPGL improves long-term outcome

SECONDARY OUTCOMES:
Time to recurrence | 18 years
  Time to recurrence
Size of recurrent tumors | 18 years
  Size of recurrent tumors
Numbers of metastases | 18 years
  Numbers of metastases
Biomarker indices of disease burden | 18 years
  Surrogate biomarker indices of disease burden (such as hormonal measures)
Metabolic parameter - blood glucose | 18 years
  fasting blood glucose
Metabolic parameter - HbA1c | 18 years
  Hb1Ac
Metabolic parameter - cholesterol | 18 years
  fasting cholesterol (total, LDL, HDL)
Hormonal parameters | 18 years
  hormonal profiles including metanephrines, normetanephrines and metoxytyramine (that will allow for sub-group specification of PPGLs)
Blood pressure profiles | 18 years
  Measurement of 24h blood pressure and ambulatory blood pressure measurments
Cardiac function | 18 years
  Leftventricualr ejection fraction
Disease specific mortality | 18 years
  Disease specific mortality
Overall mortality | 18 years
  Overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Felix Beuschlein, M.D., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided